CLINICAL TRIAL: NCT01445795
Title: A Multi-center, Placebo-controlled, Multiple Dose, Study of the Safety and Pharmacokinetics and Pharmacodynamics of INX-08189 Dosed Either QD, BID or Adjunctively With Ribavirin, and a Study of the Food Effect, in Chronically-infected Genotype 1 HCV, Treatment-naïve Subjects
Brief Title: Safety Study of INX-08189, Pharmacokinetic and Pharmacodynamic With Ribavirin and Food Effect Study, in Chronically-infected Genotype 1 Hepatitis C Virus, Treatment-naïve Subjects
Acronym: INH-189-006
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: AI472-006; INH-189-006 (Other: INH-189-006)
Record Dates: First submitted 2011-09-27; First posted 2011-10-04 (Estimated); Last update posted 2016-06-27 (Estimated); Status verified 2016-06

CONDITIONS: Hepatitis C
Keywords: Inhibitex; Chronic Hepatitis; Hepatitis C Virus
MeSH Terms: conditions — Hepatitis C; Hepatitis, Chronic | interventions — BMS-986094; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (8):
- 200 mg INX-08189 Fasted (Experimental): Cohort 1: 200 mg INX-08189 QD fasted for seven days
  Interventions: Drug: 200 mg INX-08189 Fasted
- Placebo QD Fasted (Placebo Comparator): Cohort 1: Placebo QD fasted for seven days
  Interventions: Drug: Placebo QD Fasted
- 100 mg INX-08189 with Ribavirin (Experimental): Cohort 2: 100 mg INX-08189 100 mg dosed with ribavirin x7 days (ribavirin will be dosed in a weight-based fashion as labeled BID, the AM dose will be taken 4 hours after INX-08189 so it may be taken with food)
  Interventions: Drug: 100 mg INX-08189 QD; Drug: ribavirin
- Placebo QD dosed with ribavirin (Active Comparator): Cohort 2: Placebo QD dosed with ribavirin x7 days (ribavirin will be dosed in a weight-based fashion as labeled BID)
  Interventions: Drug: Placebo QD
- 100 mg INX-08189 with a low-fat meal (Experimental): Cohort 3: 100 mg INX-08189 with a low-fat meal QD x7 days
  Interventions: Drug: 100 mg INX-08189 with low-fat meal
- Placebo with low-fat meal (Placebo Comparator): Cohort 3: Placebo administered with a low-fat meal QD for 7 days
  Interventions: Drug: Placebo with low-fat meal
- 100 mg INX-08189 Fasted (Experimental): Cohort 4: 100 mg INX-08189 BID fasted x7 days
  Interventions: Drug: 100 mg INX-08189 BID Fasted
- Placebo BID Fasted (Placebo Comparator): Cohort 4: Placebo BID fasted x7 days
  Interventions: Drug: Placebo BID Fasted

INTERVENTIONS:
Drug: 200 mg INX-08189 Fasted — 200 mg capsule INX-08189 fasted x7 days
  Arms: 200 mg INX-08189 Fasted
Drug: Placebo QD Fasted — Placebo capsule QD fasted x7 days
  Arms: Placebo QD Fasted
Drug: 100 mg INX-08189 QD — 100 mg INX-08189 capsule QD x 7 days
  Arms: 100 mg INX-08189 with Ribavirin
Drug: Placebo QD — Placebo capsule Placebo QD dosed with ribavirin x7 days (ribavirin will be dosed in a weight-based fashion as labeled BID)
  Arms: Placebo QD dosed with ribavirin
Drug: 100 mg INX-08189 with low-fat meal — INX-08189 100 mg capsule, with low-fat meal QD for seven days
  Arms: 100 mg INX-08189 with a low-fat meal
Drug: Placebo with low-fat meal — Placebo capsule administered with a low-fat meal QD for seven days
  Arms: Placebo with low-fat meal
Drug: 100 mg INX-08189 BID Fasted — 100 mg INX-08189 BID fasted x7 days
  Arms: 100 mg INX-08189 Fasted
Drug: Placebo BID Fasted — Placebo BID fasted x7 days
  Arms: Placebo BID Fasted
Drug: ribavirin
  Arms: 100 mg INX-08189 with Ribavirin

SUMMARY:
This study is to determine the safety and Pharmacokinetics (PK) and Pharmacodynamics (PD) of INH-08189 dosed once a day (QD), two times a day (BID) or adjunctively with Ribavirin and a study of the food effect in Chronically-infected Genotype 1 Hepatitis C Virus (HCV), Treatment-naïve subjects.

DETAILED DESCRIPTION:
Primary Objectives:

To evaluate in chronically-infected, non-cirrhotic, genotype 1 treatment naïve-subjects dosed with Study Drug for 7 consecutive days

Safety

- The safety of each of the 4 dosing cohorts of INX-08189 (200 mg daily (QD), 100 mg twice a day (BID), 100 mg QD with low-fat meal, and 100 mg QD with adjunctive ribavirin).

Pharmacokinetic

- To characterize the pharmacokinetic (PK) profile of oral doses of INX-08189 (200 mg QD, 100 mg BID, 100 mg QD with low-fat meal, and 100 mg QD with adjunctive ribavirin) and the PK profile of the metabolite (INX-08032).

Pharmacodynamic

- To evaluate the relationship between the kinetics of the reduction from baseline in serum HCV RNA and PK parameters of INX-08189 and the metabolite INX-08032

Efficacy

- To measure the kinetics of viral load reduction in plasma HCV RNA by each of the 4 dosing cohorts of INX-08189 (200 mg QD, 100 mg BID, 100 mg QD with low-fat meal, and 100 mg QD with adjunctive ribavirin).

ELIGIBILITY:
Inclusion Criteria:

Screening visit (Visit 1), subject criteria:

* Males and females, 18 to 65 years of age inclusive with a body mass index (BMI) of at least 18 kg/m2 but not exceeding 36 kg/m2;
* Diagnosed with chronic HCV by at least 1 previous polymerase chain reaction (PCR) result prior to Visit 1 (screening), with a positive HCV viral load of least 100,000 IU/ml at Visit 1 (screening) as measured by quantitative PCR;
* HCV genotype 1 per laboratory testing report;
* HCV treatment-naïve where "treatment-naïve" is defined as no prior treatment with interferon alpha, pegylated interferon alpha, ribavirin, or any HCV direct acting anti-viral drugs;
* Liver biopsy consistent with chronic HCV infection but with a classification of non-cirrhotic as judged by a pathologist (defined as Knodell ≤ 3, Metavir ≤ 2, Ishak ≤ 4, or Batts & Ludwig ≤ 2) within the last 2 years and before Visit 2 (biopsy can be done within the screening period);
* Negative urine drug screen for drugs of abuse (see Appendix B; note: methadone is not allowed);
* Females will have a negative serum beta human chorionic gonadotropin (βHCG) pregnancy test at screening and a negative urine dipstick pregnancy test upon entry to the clinical unit on Study Day -1;
* Agreement by both female subjects of childbearing potential and male subjects (who have not been surgically sterilized) to practice an acceptable method of birth control, which includes at least 1 barrier during the study and at least 6 months after cessation of treatment. Surgical sterilization of either the female or the male must have occurred at least 6 month prior to first dose and females must be post-menopausal for 2 years to be considered non-child-bearing potential.
* Willing and able to complete all study visits and procedures, and able to effectively communicate with the Investigator and other testing center personnel;
* Signed informed consent form (ICF) executed prior to protocol screening assessments

Exclusion Criteria:

screening visit (Visit1), subject criteria:

* Advanced liver disease, cirrhosis, or signs of decompensated liver disease such as variceal bleeding, ascites, hepatic encephalopathy, active jaundice defined by a total bilirubin > 2, or other evidence of decompensated liver disease;
* Co-infection with hepatitis B virus (HBV)or human immunodeficiency virus (HIV) (positive test for hepatitis B surface antigen [HBsAg] or anti-HIV antibody [Ab]);
* Acute cardiac ischemia, unstable heart disease or clinically symptomatic cardiac abnormalities apparent on electrocardiogram (ECG) and physical exam, or a QTcF interval at Visit 1 of ≥ 450 ms by Fridericia's correction, or a personal or family history of Torsades de pointes;
* Use of the following medications concurrently or within the 30 days prior Screening (Visit 1) associated with QT prolongation: macrolides, antiarrhythmic agents, azoles, fluoroquinolones, and tricyclic anti-depressants (note: methadone use is not allowed);
* Use of immunosuppressive or immune-modulating agents (including corticosteroids and immunosuppressive agents) or presence of an immunologically-mediated autoimmune disease (other than asthma) or history of solid organ or bone marrow transplantation (note: inhaled steroids for asthma and topical steroid for minor skin conditions allowed and washout period for PO/IM/IV corticosteroid use is 8 weeks; washout periods for other immunosuppressives determined by Medical Monitor);
* Use of strong Cytochrome P (CYP)3A4-inhibiting protease inhibitors (specifically atazanavir, indinavir, nelfinavir, saquinavir, and ritonavir), strong CYP3A4 inhibitors (specifically clarithromycin, itraconazole, ketoconazole, nefazodone, telithromycin), or strong CYP3A4 inducers (specifically rifampin, efavirenz, etravirine, phenobarbital, phenytoin, and carbamazepine);
* Absolute neutrophil count of < 1,800 cells/mm3, or platelet count < 130,000 cells/mm3, or hemoglobin < 12 g/dl for women and < 13 g/dl for men, or a history of anemia, sickle cell anemia, or thalassemia; (note: if baseline value within 5% of minimum qualifying value, 1 re-test allowed for the purpose of qualifying for study);
* A history of abnormal thyroid function that is not adequately controlled (defined as thyroid stimulating hormone [TSH] levels < 0.8 x lower limit of normal [LLN] or > 1.2 x the upper limit of normal [ULN]);
* Serum creatinine concentration ≥ 1.5 times the upper limit of normal, or albumin ≤ 3 g/dl;
* Any history of suicide attempt, receipt of professional counseling for suicidal ideation or any current suicidal ideation, or other serious psychiatric disorders (ie, bipolar disorder, severe depression, psychosis) requiring or having required hospitalization or medication
* Any malignancy within the last 5 years other than treated cervical carcinoma in situ or treated basal cell carcinoma with no more than 20% risk of recurrence within 2 years;
* Alcohol abuse within the past 2 years or an alcohol use pattern that will interfere with the study conduct;
* Drug abuse within the last 6 months.
* Current lactation or breastfeeding;
* Major surgery within 30 days prior Visit 1;
* Participation in another clinical trial of an investigational drug or device within 6 months prior to visit 1 unless that prior participation involved exposure only to placebo by clear and available documentation;
* Donation of blood or plasma within 30 days prior to Visit 1.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-09; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HCV RNA 24 hours following the final dose of Study Drug (INX-08189/placebo) | 24 hours following the final dose of Study Drug

SECONDARY OUTCOMES:
Change in HCV RNA over time during the 7 days of dosing and during the follow-up period and the maximum change from baseline in HCV RNA. | HCV RNA will be measured at the following time points: Once each at Screening (Visit1), Study Day 10 (Visit 12), and Study Day 14 (Visit 13). Samples will be taken for HCV analysis pre-dose, and at 12, 24 and 48 hours after the first dose of Study Drug

CONTACTS AND LOCATIONS:
Locations (2):
- San Antonio, Texas, United States
- San Juan, Puerto Rico